CLINICAL TRIAL: NCT07253181
Title: Tenecteplase Before inteRhospital Transfer for Endovascular Treatment in pAtientS With acUte Anterior ciRculation Large vEssel Occlusion at 4.5 to 24 Hours
Brief Title: Tenecteplase Before Interhospital Transfer for EVT in Acute Anterior Circulation LVO at 4.5-24 Hours
Acronym: TREASURE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Boehringer Ingelheim (China) Investment Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2025]372-001
Record Dates: First submitted 2025-11-13; First posted 2025-11-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke; Large Vessel Occlusion; Transportation of Patients
Keywords: interhospital transfer; acute ischemic stroke; anterior circulation large vessel occlusion
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Intervention Model Description: This is a phase Ⅲ, multicenter, prospective, randomized, open-label, blinded endpoint (PROBE) clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Except for the screening period, all endpoints will be assessed by at least on qualified blinded assessor who remains unaware of the treatment assignment. Blinded assessors must undergo a standardized training and competency validation before being delegated by the site principal investigator (PI).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tenecteplase at a nECC before EVT transfer (Experimental): Patients will receive intravenous Tenecteplase 0.25 mg/kg body-weight up to a maximum of 25mg. Transport to ECCs for EVT should be initiated as early as possible after administration.
  Interventions: Drug: Tenecteplase (TNK) (0.25 mg/kg, to maximum of 25mg)
- Direct transfer (No Intervention): Patients will be directly transferred to ECCs for EVT according to Chinese guidelines for diagnosis and treatment of acute ischemic stroke 2023.

INTERVENTIONS:
Drug: Tenecteplase (TNK) (0.25 mg/kg, to maximum of 25mg) — Tenecteplase at a nECC before EVT transfer
  Arms: Tenecteplase at a nECC before EVT transfer

SUMMARY:
This study will address the efficacy and safety of Tenecteplase administered in non-endovascular capable center (nECC) in patients with acute ischemic stroke (AIS) caused by anterior circulation large vessel occlusion (acLVO) who present in the 4.5- to 24-hour time window before interhospital transfer to a endovascular capable center (ECC) for endovascular treatment (EVT).

* Primary objective: To evaluate the efficacy of Tenecteplase administration at a nECC before EVT transfer compared with direct transfer on 90-day function outcomes;
* Secondary objective and further: To evaluate the safety of Tenecteplase administration at a nECC before EVT transfer; To evaluate the impact of time from needle-to-arterial puncture on clinical outcomes.

Patients who meet inclusion criteria will be randomized to Tenecteplase (0.25mg/kg, maximum 25mg) administered before transfer or direct transfer to ECCs. A single bolus dose should be injected over 5 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older;
* AIS symptom onset within 4.5 to 24 hours, stroke onset is defined as the time the patient was last known to be well (including wake-up stroke and unwitnessed stroke);
* Signs and symptoms consistent with the diagnosis of an acute anterior circulation ischemic stroke involving occlusion of the internal carotid artery (ICA), MCA (M1 or M2) vessels;
* Functionally independent (mRS 0-2) prior to stroke onset;
* Baseline National Institute of Health Stroke Scale (NIHSS) of 6-25;
* Intended to transfer to ECCs for EVT;
* Written informed consent from patients or legally authorized representatives;
* Neuroimaging:

  * ICA or M1, M2 occlusion by magnetic resonance angiography (MRA) or computed tomography angiography (CTA) and ANY of the following:

    1. if CT perfusion (CTP) or MR perfusion (MRP) is performed, target mismatch is defined as ischemic core volume <70mL, mismatch volume ≥15mL and mismatch ratio ≥1.8;
    2. if CTP or MRP is technically inadequate, an ASPECTS score should be of 7 or more evidenced by CT or MRI scan;

Exclusion Criteria:

* Known hypersensitivity or allergy to any ingredients of Tenecteplase;
* Rapidly improving symptoms with NIHSS score <6 before randomization;
* Any contra-indication for IVT except for the time criterion;
* Known hereditary or acquired hemorrhagic diathesis;
* Impairment in coagulation due to comorbid disease or anticoagulant use. If on warfarin, INR >1.7 or prothrombin time >15s; if use of any direct oral anticoagulant within the last 48 hours; if on any full dose heparin/heparinoid within the last 24 hours;
* Ischemic stroke or myocardial infarction in previous 3 months
* Previous intracranial hemorrhage, active internal bleeding (gastrointestinal or urinary tract hemorrhage) in previous 3 months;
* Severe, uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg);
* Other serious, advanced or terminal illness with life expectancy less than 6 months;
* Baseline blood glucose <50mg/dl or >400mg/dl;
* Contraindication to imaging with contrast agents;
* Acute symptomatic arterial occlusions in more than one vascular territory confirmed on CTA or MRA (e.g. bilateral MCA occlusions, or an MCA and a basilar artery occlusion);
* Extensive early ischemic change on non-contrast CT estimated to be >1/3 MCA territory, or significant hypodensity outside the Tmax>6s perfusion lesion that invalidates mismatch criteria;
* Evidence of intracranial tumor (mass effect), acute intracranial hemorrhage, or arteriovenous malformation;
* Current participation in another investigational drug or device study;
* Suspected endocarditis;
* Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Ordinal mRS score | at 90 (±7) days
  the ordinal score on the modified Rankin scale; The modified Rankin scale is a measure of disability, with scores ranging from 0 (no symptoms) to 6 (death).

SECONDARY OUTCOMES:
Dichotomized mRS of 0-1 vs. 2-6 | at 90 (±7) days
Dichotomized mRS of 0-2 vs. 3-6 | at 90 (±7) days
Dichotomized mRS of 0-3 vs. 4-6 | at 90 (±7) days
Score on the EQ-5D-5L | at 90 (±7) days
  Health-related quality of life (the score on the EuroQol Group 5-Dimension 5-Level [EQ-5D-5L] questionnaire; range, -0.39 to 1, with higher scores indicating better quality of life)
Incidence of arterial recanalization | Day 1
  Arterial imaging performed at ECC arrival, either CTA/MRA/or first run of DSA
Recanalization | at 24 (±12) hours
First pass reperfusion | intraoperative, immediately after the first pass
  First pass reperfusion refers to achievement of recanalization by single pass, near-complete to complete recanalization of the occlusion site (eTICI 2c or 3) and no need for rescue treatment
Successful reperfusion | immediately after the endovascular intervention
  successful reperfusion is defined as extended Treatment In Cerebral Ischemia (eTICI) grades of 2b, 2c or 3

OTHER OUTCOMES:
Symptomatic intracranial hemorrhage (sICH) | within 36 hours
  using Heidelberg criteria
Parenchymal hematoma type 2 (PH2) | within 36 hours
All-cause mortality | up to 90 (±7) days
Change in Infarct volume | Day 1
  Measured by neuro imaging at baseline and ECC arrival
Hemorrhagic transformation | Day 1
  Measured by neuro imaging at ECC arrival

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, MD, PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (2):
- China (2):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Affiliated Hospital of Shandong Second Medical University, Weifang, Shandong

IPD SHARING:
Plan to Share IPD: No
According to Chinese laws and regulations, the IPD will not be shared.